CLINICAL TRIAL: NCT05117190
Title: Human Composite Facial Allotransplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 028.TRN.2014.D
Record Dates: First submitted 2015-04-15; First posted 2021-11-11 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Transplantation: Facial Transplantation
Keywords: Facial Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Facial Deformity (Other): Face not the normal shape because of injury or illness.
  Interventions: Procedure: Facial Allotransplantation

INTERVENTIONS:
Procedure: Facial Allotransplantation

SUMMARY:
Allotransplantation of maxillofacial of subject with severe facial deformities due to traumatic events.

DETAILED DESCRIPTION:
A facial transplantation is a highly dynamic, prolonged operation requiring teams communicating seamlessly through its duration. This is similar to complex solid organ transplant teams at Methodist Transplant Institute. The Institute's clinical experience in management of complex facial defects and deformities along with the personnel and infrastructure at Methodist Dallas transplant institute would help develop a center for Facial Allotransplantation. The team experience, true collaboration, creativity and a unique approach to each patient would help provide the optimal care and reconstruction for the face allotransplant patient both before and after surgery.

The purpose of this study is centered on the advancement of a safe and effective procedure for Facial Allotransplantation at Methodist Hospital Medical Center at Dallas. Composite tissue allotransplantation for facial reconstruction is in its infancy as liver transplantation was 30 years ago when the first liver transplant was completed in Texas. This study will establish Methodist Hospital System as a center for Facial Allotransplantation for reconstruction of extensive facial defects resulting in functional loss and poor quality of life.

Patient participation post transplantation will either be for life, or failure of the composite tissue allograft. Patient enrollment will be initiated immediately after the IRB approval. The enrollment period will be completed after the patient receives the final transplant, and the study will be completed at 24 months after the final transplant. However, all patients enrolled into the study will have lifelong follow up with immunosuppressive management, psychological support, and evaluation of functional recovery per protocol.

ELIGIBILITY:
Inclusion Criteria:

* Between ages 18-70 years
* Must be willing to undergo major facial reconstruction
* Be able to understand the pre and post-transplantation evaluation, physical therapy, and follow up procedures
* Conventional reconstruction deemed unsatisfactory

Exclusion Criteria:

* Medically unable to provide consent
* Active infections such as Human Immunodeficiency Virus, mycobacteria, hepatitis B, and hepatitis C
* Recent history of alcohol or IV drug or chemical dependency
* Psychiatric evaluation that indicate mental instability or non-compliance
* Cognitively impaired and Terminally ill
* Women of child bearing age with intent to conceive, pregnant or lactating
* Unable to receive immunosuppression after transplantation because of either geographic or financial limitations
* End stage organ disease (renal failure, Congestive Heart Failure (CHF), Chronic Obstructive Pulmonary Disease (COPD), etc.)
* Chronic infections such as osteomyelitis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-10-21 (Actual); Primary Completion 2021-03-18 (Actual); Study Completion 2021-03-18 (Actual)

PRIMARY OUTCOMES:
Modified Facial Clinimetric Evaluation Scale | measured at 6 weeks
  validated quality-of-life instrument that is used to assess facial impairment and disability after facial paralysis.
Modified Facial Clinimetric Evaluation Scale | measured at 3 months
  validated quality-of-life instrument that is used to assess facial impairment and disability after facial paralysis.
Modified Facial Clinimetric Evaluation Scale | measured at 6 months
  validated quality-of-life instrument that is used to assess facial impairment and disability after facial paralysis.
Modified Facial Clinimetric Evaluation Scale | measured at 12 months
  validated quality-of-life instrument that is used to assess facial impairment and disability after facial paralysis.
Modified Facial Clinimetric Evaluation Scale | measured at 18 months
  validated quality-of-life instrument that is used to assess facial impairment and disability after facial paralysis.
Modified Facial Clinimetric Evaluation Scale | measured at 24 months
  validated quality-of-life instrument that is used to assess facial impairment and disability after facial paralysis.
Facial Disability Index | measured at 6 weeks
  a disease-specific, self-report instrument for the assessment of disabilities of patients with facial nerve disorders
Facial Disability Index | measured at 3 months
  a disease-specific, self-report instrument for the assessment of disabilities of patients with facial nerve disorders
Facial Disability Index | measured at 6 months
  a disease-specific, self-report instrument for the assessment of disabilities of patients with facial nerve disorders
Facial Disability Index | measured at 12 months
  a disease-specific, self-report instrument for the assessment of disabilities of patients with facial nerve disorders
Facial Disability Index | measured at 18 months
  a disease-specific, self-report instrument for the assessment of disabilities of patients with facial nerve disorders
Facial Disability Index | measured at 24 months
  a disease-specific, self-report instrument for the assessment of disabilities of patients with facial nerve disorders
SF-36 Health Survey | measured at 6 weeks
  a set of generic, coherent, and easily administered quality-of-life measures
SF-36 Health Survey | measured at 3 months
  a set of generic, coherent, and easily administered quality-of-life measures
SF-36 Health Survey | measured at 6 months
  a set of generic, coherent, and easily administered quality-of-life measures
SF-36 Health Survey | measured at 12 months
  a set of generic, coherent, and easily administered quality-of-life measures
SF-36 Health Survey | measured at 18 months
  a set of generic, coherent, and easily administered quality-of-life measures
SF-36 Health Survey | measured at 24 months
  a set of generic, coherent, and easily administered quality-of-life measures

CONTACTS AND LOCATIONS:
Overall Officials: Likith V. Reddy, MD, Principal Investigator — Methodist Health System
Locations (1):
- Methodist Health System, Dallas, Texas, United States